CLINICAL TRIAL: NCT06254079
Title: The Effect of Video-based Training Given by Operating Room Nurses to Patients Undergoing Laparoscopic Cholecystectomy on Anxiety, Pain and Recovery Quality.
Brief Title: The Effect of Video-based Education on Anxiety, Pain and Recovery Quality in Patients Undergoing Laparoscopic Cholecystectomy.
Acronym: EDUCATION
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Yeliz Sürme, Principal Investigator, Assoc.Prof. Dr, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2023/46
Record Dates: First submitted 2024-01-31; First posted 2024-02-12 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Laparoscopic Cholecystectomy
Keywords: Video-based education; Operating room nurse; Laparoscopic Cholecystectomy

STUDY DESIGN:
Intervention Model Description: designed as a randomized controlled experimental
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): A video containing information about the operating room environment and intraoperative care will be watched. The patients who watch the video will be questioned again about the points they do not understand, the issues they are curious about about the perioperative period, and the information they want to learn, and this information will be given verbally by the researchers.
  Interventions: Procedure: video based education
- Control Group (No Intervention): Patients in this group will not be shown any videos and will continue to receive care according to their clinical routine.They will be asked to answer the questions in the patient introduction form the day before the surgical intervention. The surgical anxiety scale will be filled in when patients come from the ward to the preoperative waiting room on the day of surgery. Finally, patients will be asked to answer the questions on VAS and Quality of Recovery-15 (QoR-15) in the patient room at the 24th hour after surgery.

INTERVENTIONS:
Procedure: video based education — The patients in the experimental group will be shown a video containing information about the operating room environment and care during surgery. The video content includes the following details: the operating room temperature being maintained at 18-24°C; the patient being placed on the operating table by the staff in the presence of an anesthesia technician; the establishment of intravenous access by the anesthesia technician; monitoring of blood pressure, pulse, respiration, and EKG indicators; the insertion of a urinary catheter by the surgical nurse after the patient is anesthetized; post-awakening transfer to the postoperative recovery unit with the anesthesia technician and personnel; reception and monitoring of vital signs, pain assessment, intervention, and observation for a period by a nurse in this unit; and finally, transfer to the General Surgery Service.
  Arms: Intervention group

SUMMARY:
The reasons for anxiety before laparoscopic cholecystectomy include the operation of the surgery process, its therapeutic effect, lack of information about the postoperative period and lack of communication. The increase in the preoperative anxiety level in patients undergoing surgical intervention negatively affects the patients' sleep, recovery and quality of life, length of hospital stay is prolonged, cost increases in hospitals, and socioeconomic losses occur in individuals and institutions. Therefore, this study will be conducted as a randomized controlled experimental study to determine the effect of video-based training given by an operating room nurse to patients undergoing laparoscopic cholecystectomy on preoperative anxiety, postoperative pain and recovery quality.

Considering possible sample loss, it was decided to include 72 patients, 36 in the intervention group and 36 in the control group. One of the patients included in both the intervention and control groups was excluded from the study because he was converted to open cholecystectomy during surgery and was taken to intensive care postoperatively. The study was completed with a total of 70 patients, 35 in the intervention group and 35 in the control group.

Patient Information Form, Surgical Anxiety Scale, Visual Analogue Scale (VAS) and Recovery Quality Scale-15 will be used to collect data.

DETAILED DESCRIPTION:
A total of 2 patients, 1 patients in the experimental and 1 patients in the control groups, were excluded from the study because they were converted from laparoscopic surgery to open surgery.The study was completed with 70 patients (35 experimental and 35 control) who underwent laparoscopic cholecystectomy and met the inclusion criteria.

ELIGIBILITY:
Inclusion Criteria:

* Agreeing to participate in the research,

  * Knows how to read, write and speak Turkish,
  * Patients who will undergo elective laparoscopic cholecystectomy in the General Surgery Service will be included.

Exclusion Criteria:

* Have cognitive, auditory and psychological problems that may affect communication with researchers,
* Using psychiatric medication,
* Undergoing surgical intervention under emergency conditions,
* Subjected to spinal, epidural or local anesthesia during surge

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Video based education | 1 day
  The video includes information about various aspects such as preoperative waiting and postoperative recovery units, the operating room, tables with surgical instruments, sterile drapes, and characteristics of surgical team members. Additionally, details are provided regarding the information to be obtained from patients upon arrival in the operating room, positions to be instructed for the surgical procedure and corresponding precautions, communication methods with the patient's family during the surgery, interventions in the postoperative recovery unit, and criteria for transferring patients to the regular service after surgery.

SECONDARY OUTCOMES:
Surgical Anxiety | 1 day
  The surgical anxiety scale will be filled out when patients come from the ward to the preoperative waiting room on the day of surgery.Scores between 0 and 60 are taken from the scale. As the score obtained from the scale increases, the individual's anxiety is interpreted as high.
Visual Analog Scale Pain | up to 24 hours
  Application of visual analog scale pain to all patients at the 24 hours later after surgery. The range of scores on the scale varies between 0-10, and higher scores indicate increased pain intensity.
Recovery Quality | up to 24 hours
  The Quality of Healing-15 Scale was completed by all patients 24 hours later after the surgery.The score range that can be obtained from the scale varies between 0-150. As the score increases, the quality of recovery increases.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Erciyes University, Kayseri, Talas
  - Erciyes University, Kayseri

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Stark PA, Myles PS, Burke JA. Development and psychometric evaluation of a postoperative quality of recovery score: the QoR-15. Anesthesiology. 2013 Jun;118(6):1332-40. doi: 10.1097/ALN.0b013e318289b84b. PMID 23411725
- [Result] Dolan R, Huh J, Tiwari N, Sproat T, Camilleri-Brennan J. A prospective analysis of sleep deprivation and disturbance in surgical patients. Ann Med Surg (Lond). 2016 Jan 6;6:1-5. doi: 10.1016/j.amsu.2015.12.046. eCollection 2016 Mar. PMID 26909151
- [Result] Gursoy A, Candas B, Guner S, Yilmaz S. Preoperative Stress: An Operating Room Nurse Intervention Assessment. J Perianesth Nurs. 2016 Dec;31(6):495-503. doi: 10.1016/j.jopan.2015.08.011. Epub 2016 May 6. PMID 27931701